CLINICAL TRIAL: NCT02625974
Title: Prospective, Historically Controlled Study to Evaluate the Efficacy and Safety of a New Pediatric Formulation of Nifurtimox in Children Aged 0 to 17 Years With Chagas' Disease
Brief Title: A Study to Learn How Well Nifurtimox Works and How Safe it is in Children Aged 0 to 17 Years With Chagas' Disease, an Inflammatory, Infectious Disease Caused by the Parasite Trypanosoma Cruzi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16027; 2022-001504-17 (EudraCT Number)
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Chagas Disease
MeSH Terms: conditions — Chagas Disease | interventions — Nifurtimox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Nifurtimox 60 days / Arm 1 (Experimental): Nifurtimox tablets administered three times daily for 60 days (Days 1 - 60, active nifurtimox treatment)
  Interventions: Drug: Nifurtimox (Lampit, BAYA2502)
- Nifurtimox 30 days / Arm 2 (Experimental): Nifurtimox tablets administered three times daily for 30 days, followed by placebo administered three times daily for 30 days (Days 1 - 30, active nifurtimox treatment; Days 31 - 60, placebo)
  Interventions: Drug: Nifurtimox (Lampit, BAYA2502); Drug: Placebo

INTERVENTIONS:
Drug: Nifurtimox (Lampit, BAYA2502) — For pediatric participants with body weight ≤ 40 kg: dosage 10 to 20 mg/kg/day in three divided doses.
  For pediatric participants with body weight > 40 kg: 8 - 10 mg/kg/day in three divided doses.
  60 days or 30 days of nifurtimox treatment
Drug: Placebo — Matching placebo
  Arms: Nifurtimox 30 days / Arm 2

SUMMARY:
Researchers are looking for a better way to treat children who have an infectious disease caused by the parasite Trypanosoma cruzi (Chagas' disease).

Chagas'disease is an inflammatory, infectious disease caused by the parasite Trypanosoma cruzi. This parasite is mainly spread by insects called triatomine bug. If Chagas' disease is left untreated, it can later cause serious heart and digestive problems.

The study treatment nifurtimox has been used for more than 50 years to treat Chagas' disease. When used early after infection, it kills the parasite. In people who have long-term Chagas' disease, it's no longer possible to kill the parasite. However, nifurtimox may help slow the progression of the disease and its most serious complications.

Nifurtimox was developed for use in adults only, but has also been used in children (off-label) for over 40 years. Currently it is available for doctors to give to adults and to children. However, there are not enough data about nifurtimox in children.

The main purpose of this study is to learn how well nifurtimox works in children aged 8 months to less than 18 years with Chagas' disease. To answer this, the researchers will compare the amount of antibodies against the parasite Trypanosoma cruzi in the serum (fluid from blood without the clotting factors) between children treated with nifurtimox for 60 days with untreated children from the past (control group):

* 12 months and
* 4 years after the end of treatment. The data for the control group will come from 2 previous studies conducted in children.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Male and female pediatric subjects aged 0 days to younger than 18 years
* Chagas' disease diagnosed/ confirmed for a) Subjects < 8 months of age at randomization must demonstrate direct observation of Trypanosoma cruzi by concentration test; b) Subjects ≥ 8 months to < 18 years of age at randomization must demonstrate a positive conventional ELISA result for both recombinant ELISA and total purified antigen ELISA

Part 2:

- Male and female subjects who were randomized and received at least one dose of their assigned 60- or 30-day regimen of nifurtimox treatment

Exclusion Criteria:

Part 1:

* Subjects aged 0 to 27 days who, at birth, were pre-term, weighed less than 2500 g, or had a maximum Apgar score < 7 at 5 minutes
* Known evidence of Chagas' disease-related cardiomyopathy/ Chagas' heart disease
* Known evidence of Chagas' disease-related gastrointestinal dysfunction (e.g. megaoesophagus, megacolon, or both) or Chagas' digestive disease
* Serious manifestations of acute Chagas' disease, including myocarditis, meningoencephalitis, or pneumonitis
* Known evidence of Chagas' disease-related damage to the peripheral nervous system or peripheral neuropathy
* Clinically significant psychiatric disorder (e.g. moderate to severe depression, severe anxiety, or psychosis) or epilepsy
* Subjects with contraindications/ warnings to nifurtimox administration, or with conditions that may increase the risk of the undesirable effects of nifurtimox
* Subjects who have had previous treatment with trypanocidal agents or an accepted indication for antiparasitic therapy (e.g. reactivation of Chagas' infection due to immunosuppression by several diseases or treatment with steroids)
* Subjects living in housing conditions where there is no active or effective vector control to Trypanosoma cruzi reinfection as determined by Ministry of Health guidelines in each country

Part 2:

* Subjects with acute or chronic health conditions or congenital disorders which, in the opinion of the investigator, would make them unsuitable for participation in the clinical study
* Subjects living in housing conditions where there is no active or effective vector-control to Trypanosoma cruzi reinfection as determined by Ministry of Health guideline of the respective country
* Subjects with clinical manifestations of Chagas' disease-related gastrointestinal dysfunction or serious manifestations of acute Chagas' disease
* Immuno-compromised subjects (e.g. with human immunodeficiency virus or treated with immunosuppressive drugs)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Argentina (13):
  - La Plata, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - San Salvador de Jujuy, Jujuy Province
  - Posadas, Misiones Province
  - Rosario, Santa Fe Province
  - Corrientes
  - Formosa
  - La Rioja
  - Mendoza
  - Salta
  - San Juan
  - San Miguel de Tucumán
  - Santiago del Estero
- Bolivia (3):
  - Cochabamba
  - Punata
  - Tarija
- Colombia (4):
  - Soledad, Atlántico
  - Yopal, Casanare Department
  - Santa Marta, Magdalena Department
  - Floridablabca, Santander Department

REFERENCES:
- [Result] Sosa Estani S, Segura EL, Ruiz AM, Velazquez E, Porcel BM, Yampotis C. Efficacy of chemotherapy with benznidazole in children in the indeterminate phase of Chagas' disease. Am J Trop Med Hyg. 1998 Oct;59(4):526-9. doi: 10.4269/ajtmh.1998.59.526. PMID 9790423
- [Result] de Andrade AL, Zicker F, de Oliveira RM, Almeida Silva S, Luquetti A, Travassos LR, Almeida IC, de Andrade SS, de Andrade JG, Martelli CM. Randomised trial of efficacy of benznidazole in treatment of early Trypanosoma cruzi infection. Lancet. 1996 Nov 23;348(9039):1407-13. doi: 10.1016/s0140-6736(96)04128-1. PMID 8937280
- [Result] Altcheh J, Castro L, Dib JC, Grossmann U, Huang E, Moscatelli G, Pinto Rocha JJ, Ramirez TE; CHICO Study Group. Prospective, historically controlled study to evaluate the efficacy and safety of a new paediatric formulation of nifurtimox in children aged 0 to 17 years with Chagas disease one year after treatment (CHICO). PLoS Negl Trop Dis. 2021 Jan 7;15(1):e0008912. doi: 10.1371/journal.pntd.0008912. eCollection 2021 Jan. PMID 33412557
- [Derived] Rivero R, Esteva MI, Huang E, Colmegna L, Altcheh J, Grossmann U, Ruiz AM; CHICO and CHICO SECURE Study Groups. ELISA F29 -A therapeutic efficacy biomarker in Chagas disease: Evaluation in pediatric patients treated with nifurtimox and followed for 4 years post-treatment. PLoS Negl Trop Dis. 2023 Jun 23;17(6):e0011440. doi: 10.1371/journal.pntd.0011440. eCollection 2023 Jun. PMID 37352322
- [Derived] Altcheh J, Sierra V, Ramirez T, Pinto Rocha JJ, Grossmann U, Huang E, Moscatelli G, Ding O. Efficacy and Safety of Nifurtimox in Pediatric Patients with Chagas Disease: Results at 4-Year Follow-Up in a Prospective, Historically Controlled Study (CHICO SECURE). Antimicrob Agents Chemother. 2023 Apr 18;67(4):e0119322. doi: 10.1128/aac.01193-22. Epub 2023 Mar 28. PMID 36975790
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=16027&attachmentIdentifier=341adaa4-a747-4150-98c6-4f09a62e7bcb&fileName=Bayer_16027_PLS_v2.0_2022_08_30.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 of the study was conducted from 27 JAN 2016 (First subject first visit) to 25 JUL 2018 (Last subject last visit) in Argentina, Bolivia and Colombia.
  Part 2 of the study was conducted from 26 SEP 2018 (First subject first visit) to 10 AUG 2021 (Last subject last visit) in Argentina, Bolivia and Colombia.
Pre-assignment Details: Part 1: 330 subjects who were eligible to participate in the study were randomized in a 2:1 ratio to either a 60-Day or 30-Day regimen with nifurtimox tablets. 308 subjects completed treatment in Part 1, and 318 subjects completed Part 1.
  Part 2: Of the 318 subjects completed Part 1, 295 subjects were included in Part 2.
Groups:
- Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2: Nifurtimox tablets administered three times daily for 30 days, followed by placebo administered three times daily for 30 days (Days 1 - 30, active nifurtimox treatment; Days 31 - 60, placebo)
Period: Part 1
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Started | 219 | 111
Received Treatment | 219 | 111
Completed | 210 | 108
Not Completed | 9 | 3
Not completed — Lost to Follow-up | 9 | 3
Period: Part 2
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Started | 197 | 98
Completed | 191 | 91
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 4 | 6
Not completed — Other, including due to the COVID-19 Pandemic | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2 | Nifurtimox 60 Days / Arm 1 | Total
Number analyzed (Participants) | 111 | 219 | 330
Age, Customized [Count of Participants; unit: Participants]
  0 to 27 days | 3 | 4 | 7
  28 days to younger than 8 months | 4 | 8 | 12
  8 months to younger than 2 years | 8 | 17 | 25
  2 years to younger than 18 years | 96 | 190 | 286
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 119 | 178
  Male | 52 | 100 | 152
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 81 | 155 | 236
  American Indian or Alaska native | 30 | 64 | 94
Total Purified Antigen enzyme-linked immunosorbent assay (ELISA) test results [Count of Participants; unit: Participants] — Chagas disease diagnosed by direct observation of T. cruzi by concentration test (subjects <8 months of age at randomization) or positive conventional ELISA results for both recombinant ELISA and total purified antigen ELISA (subjects ≥8 months to younger than 18 years of age at randomization) as determined by local laboratory test results were eligible for enrollment.
  Participants
    Reactive | 110 | 219 | 329
    Non Reactive | 1 | 0 | 1
Total Purified Antigen ELISA optical density (OD) values [Mean (Standard Deviation); unit: No dimension] | 1.532 (0.533) | 1.474 (0.553) | 1.494 (0.546)
Recombinant ELISA test results [Count of Participants; unit: Participants] — Chagas disease diagnosed by direct observation of T. cruzi by concentration test (subjects <8 months of age at randomization) or positive conventional ELISA results for both recombinant ELISA and total purified antigen ELISA (subjects ≥8 months to younger than 18 years of age at randomization) as determined by local laboratory test results were eligible for enrollment.
  Participants
    Reactive | 110 | 219 | 329
    Non Reactive | 1 | 0 | 1
Recombinant ELISA OD values [Mean (Standard Deviation); unit: No dimension] | 2.765 (0.605) | 2.735 (0.640) | 2.745 (0.628)
Non conventional ELISA-F29 test results [Count of Participants; unit: Participants] — The non-conventional ELISA-F29 test is considered an early marker of treatment efficacy in chronic Chagas disease.
  Participants
    Reactive | 72 | 142 | 214
    Non Reactive | 39 | 77 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 108 | 217 | 325
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Concentration test for T. cruzi [Count of Participants; unit: Participants] — Chagas disease diagnosed by direct observation of T. cruzi by concentration test (subjects <8 months of age at randomization).
  Participants
    Positive | 7 | 12 | 19
    Negative | 0 | 0 | 0
    Missing | 104 | 207 | 311

OUTCOME MEASURES:

1. Primary Outcome: Part 1 - Percentage of Sero-reduction or Sero-conversion (Cured Subjects)
Description: Cure is defined as sero-reduction (in subjects ≥8 months to <18 years of age at randomization) or sero-conversion (in all subjects). Sero-reduction is defined as a ≥20% reduction in optical density [OD]) measured by two conventional ELISA serology tests and sero-conversion is defined as negative Immunoglobulin G (IgG) concentration measured by two conventional ELISA serology tests.
  Subjects who have missing conventional serology results at the 12 month time point were treated as failures (ie, no cure).
  For the primary objective in the study, superiority over placebo was confirmed if the lower limit of the 95% Confidence Interval (CI) for the nifurtimox (60-day regimen) cure rate is greater than 16%, the larger of the upper limits of the 95% CIs for historical placebo control.
Time Frame: At 12 months post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Percentage of subjects | 32.9 [26.4 to 39.3] | 18.9 [11.2 to 26.7]
Statistical Analysis 1: Comparison: Nifurtimox 60 Days / Arm 1 vs Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2; Test type: Other — A direct comparison; Difference in cure rate = 14, 95% CI 2-sided [3.7 to 24.2]

2. Primary Outcome: Part 2 - Incidence Rate of Seronegative Conversion in Subjects Received at Least One Dose of the 60-day Nifurtimox Treatment Regimen.
Description: Seronegative conversion measured by two types of assay (recombinant ELISA and indirect hemagglutination assay [IHA]) in subjects who were randomized and received at least one dose of the 60-day nifurtimox treatment regimen compared to an external control group of historical placebo patients with Chagas' disease. Incidence rate is the number of new cases of seronegative conversion over the study period (i.e., 4 years after end of nifurtimox treatment) divided by the person-time at risk. It was modelled using a Poisson distribution with a 2-sided 95% exact CI.
  Number of participants with events were reported.
Time Frame: Subjects participating in Part 2 were followed up for another 3 years, for a total follow-up period of 4 years after end of nifurtimox treatment in Part 1
Measure: Number; unit: Participants
Groups:
- Nifurtimox 60 Days / Arm 1: Nifurtimox tablets administered three times daily for 60 days (Days 1 - 60, active nifurtimox treatment)
  Treatment administered in Part 1; no study drug was administered in Part 2
Arm/Group | Nifurtimox 60 Days / Arm 1
Number analyzed (Participants) | 197
Participants | 16
Statistical Analysis 1: Comparison: Nifurtimox 60 Days / Arm 1; Test type: Other — Incidence rate and 95% CI of seronegative conversion; Risk Ratio (RR) = 2.12, 95% CI 2-sided [1.21 to 3.45] — Person-year = 754

3. Secondary Outcome: Part 1 - Nifurtimox Concentration Over Time in Plasma at Visit 2
Description: Measured in sub-population.
Time Frame: At Visit 2 (Day 1): Pre-dose and Post-dose at 5-10 minutes, 10-120 minutes, 2-4 hours, and 4-8 hours
Measure: Median (Full Range); unit: ug/L
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 40 | 23
ug/L
  Predose | NA [NA to 26.8] — below the level of detection | NA [NA to NA] — below the level of detection
  5 - 10 MIN POST | NA [NA to 154.8] — below the level of detection | 21.1 [NA to 695.0] — below the level of detection
  10 - 120 MIN POST | 78.2 [5.8 to 847.5] | 49.0 [NA to 524.3] — below the level of detection
  2 - 4 HOURS POST | 215.4 [77.9 to 516.3] | 300.7 [106.9 to 533.5]
  4 - 8 HOURS POST | 267.6 [40.2 to 508.1] | 289.6 [103.2 to 301.0]

4. Secondary Outcome: Part 1 - Nifurtimox Concentration Over Time in Plasma at Visit 3
Description: Measured in sub-population.
Time Frame: At Visit 3 (Day 7): Pre-dose and Post-dose at 5-10 minutes, 10-120 minutes, 2-4 hours, and 4-8 hours
Measure: Median (Full Range); unit: ug/L
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 40 | 22
ug/L
  Predose | 47.7 [NA to 407.6] — below the level of detection | 38.3 [NA to 472.3] — below the level of detection
  5 - 10 MIN POST | 82.6 [NA to 561.6] — below the level of detection | 56.0 [NA to 442.8] — below the level of detection
  10 - 120 MIN POST | 250.6 [13.8 to 1035.6] | 232.3 [13.9 to 706.3]
  2 - 4 HOURS POST | 497.2 [57.1 to 1027.4] | 257.7 [46.3 to 660.2]
  4 - 8 HOURS POST | 427.5 [141.2 to 778.2] | 267.0 [NA to 339.6] — below the level of detection

5. Secondary Outcome: Part 1 - Nifurtimox Concentration Over Time in Plasma at Visit 6
Description: The evaluation was based on clinical examinations. Measured in sub-population.
Time Frame: At Visit 6 (Day 30): Pre-dose and Post-dose at 5-10 minutes, 10-120 minutes, 2-4 hours, and 4-8 hours
Measure: Median (Full Range); unit: ug/L
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 35 | 24
ug/L
  Predose | 23.8 [NA to 459.3] — below the level of detection | 40.8 [NA to 284.3] — below the level of detection
  5 - 10 MIN POST | 71.7 [NA to 153.7] — below the level of detection | 73.7 [NA to 266.7] — below the level of detection
  10 - 120 MIN POST | 135.0 [NA to 932.4] — below the level of detection | 172.7 [14.1 to 387.3]
  2 - 4 HOURS POST | 369.5 [92.1 to 1277.0] | 103.8 [12.3 to 1107.2]
  4 - 8 HOURS POST | 249.7 [70.9 to 504.3] | 165.2 [84.9 to 1089.3]

6. Secondary Outcome: Part 1 - Nifurtimox Concentration Over Time in Plasma at Visit 8
Description: Measured in sub-population.
Time Frame: At Visit 8 (Day 60): Pre-dose and Post-dose at 5-10 minutes, 10-120 minutes, 2-4 hours, and 4-8 hours
Measure: Median (Full Range); unit: ug/L
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 36 | 19
ug/L
  Predose | NA [NA to 258.7] — below the level of detection | NA [NA to NA] — below the level of detection
  5 - 10 MIN POST | 92.4 [15.9 to 255.1] | NA [NA to NA] — below the level of detection
  10 - 120 MIN POST | 139.1 [23.6 to 711.4] | NA [NA to 21.5] — below the level of detection
  2 - 4 HOURS POST | 395.6 [166.9 to 883.0] | NA [NA to NA] — below the level of detection
  4 - 8 HOURS POST | 300.6 [28.5 to 1217.2] | NA [NA to NA] — below the level of detection

7. Secondary Outcome: Part 2 - Incidence Rate of Seronegative Conversion in Subjects Who Received at Least One Dose of the 30-day Nifurtimox Treatment Regimen
Description: Seronegative conversion measured by two types of assay (recombinant ELISA and indirect hemagglutination assay [IHA]) in subjects who were randomized and received at least one dose of the 30-day nifurtimox treatment regimen. Incidence rate is the number of new cases of seronegative conversion over the study period (i.e., 4 years after end of nifurtimox treatment) divided by the person-time at risk. It was modelled using a Poisson distribution with a 2-sided 95% exact CI.
  Number of participants with events were reported.
Time Frame: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2: Nifurtimox tablets administered three times daily for 30 days, followed by placebo administered three times daily for 30 days (Days 1 - 30, active nifurtimox treatment; Days 31 - 60, placebo)
  Treatment administered in Part 1; no study drug was administered in Part 2
Arm/Group | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 98
Participants | 8
Statistical Analysis 1: Comparison: Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2; Test type: Other — Incidence rate and 95% CI of seronegative conversion; Risk Ratio (RR) = 2.11, 95% CI 2-sided [0.91 to 4.16] — Person-year = 379

8. Secondary Outcome: Part 2 - ECG Signs of Established Chagas-related Cardiomyopathy
Description: Summary of subjects by evidence of established Chagas-related cardiomyopathy as measured by electrocardiogram (ECG).
  Evidence of established Chagas-related cardiomyopathy: Total
Time Frame: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Nifurtimox 60 Days: Chagas-related Cardiomyopathy; Nifurtimox 30 Days: Chagas-related Cardiomyopathy: ECG signs
Arm/Group | Nifurtimox 60 Days: Chagas-related Cardiomyopathy | Nifurtimox 30 Days: Chagas-related Cardiomyopathy
Number analyzed (Participants) | 197 | 98
Participants
  YES | 0 | 0
  NO | 189 | 90
  MISSING | 8 | 8

9. Secondary Outcome: Part 2 - Serological Response of Established Chagas-related Cardiomyopathy
Description: Summary of subjects by evidence of established Chagas-related cardiomyopathy as measured by Serological response.
  Evidence of established Chagas-related cardiomyopathy: Total
Time Frame: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Nifurtimox 60 Days: Chagas-related Cardiomyopathy; Nifurtimox 30 Days: Chagas-related Cardiomyopathy: Serological response
Arm/Group | Nifurtimox 60 Days: Chagas-related Cardiomyopathy | Nifurtimox 30 Days: Chagas-related Cardiomyopathy
Number analyzed (Participants) | 197 | 98
Participants
  Non Reactive | 14 | 6
  Reactive | 176 | 84
  Missing | 7 | 8

10. Secondary Outcome: Part 1 + Part 2 - Serial Reduction of Optical Density Values Measured by Total Purified Antigen ELISA
Description: Summary and change from baseline of optical density values measured by total purified antigen ELISA.
  Optical density is the measure of absorbance, and is defined as the ratio of the intensity of light falling upon a material and the intensity transmitted.
Time Frame: Baseline and Subjects participating in Part 2 were followed up for another 3 years, for a total follow-up period of 4 years after end of nifurtimox treatment in Part 1
Measure: Mean (Standard Deviation); unit: Optical density
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 197 | 98
Optical density
  Part 1 - Baseline (Visit 1) | 1.47 (0.55) [0.55 to 2.6] | 1.52 (0.55) [lower limit 0.55]
  Part 1 - Up to 420 days post-treatment (Visit 11) | 1.24 (0.62) [0.62 to 2.5] | 1.30 (0.61) [lower limit 0.61]
  Part 1 - Change from Baseline (Visit 11) | -0.24 (0.29) [0.29 to 0.3] | -0.23 (0.41) [lower limit 0.41]
  Part 2 - Year 2: (FU Visit 1) | 1.23 (0.59) [lower limit 0.59] | 1.29 (0.61) [lower limit 0.61]
  Part 2 - Year 2: Change from Baseline (FU Visit 1) | -0.25 (0.41) [lower limit 0.41] | -0.23 (0.49) [lower limit 0.49]
  Part 2 - Year 3 (FU Visit 3) | 1.16 (0.58) [lower limit 0.58] | 1.23 (0.58) [lower limit 0.58]
  Part 2 - Year 3: Change from Baseline (FU Visit 3) | -0.30 (0.42) [lower limit 0.42] | -0.30 (0.50) [lower limit 0.50]
  Part 2 - Year 4 (FU Visit 5) | 1.12 (0.57) [lower limit 0.57] | 1.23 (0.59) [lower limit 0.59]
  Part 2 - Year 4: Change from Baseline (FU Visit 5) | -0.35 (0.40) [lower limit 0.40] | -0.30 (0.46) [lower limit 0.46]

11. Secondary Outcome: Part 1 + Part 2 - Serial Reduction of Optical Density Values Measured by Recombinant ELISA
Description: Summary and change from baseline of optical density values measured by recombinant ELISA.
  Optical density is the measure of absorbance, and is defined as the ratio of the intensity of light falling upon a material and the intensity transmitted.
Time Frame: as for outcome 10
Measure: Mean (Standard Deviation); unit: Optical density
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 197 | 98
Optical density
  Part 1 - Baseline (Visit 1) | 2.74 (0.63) [lower limit 0.63] | 2.73 (0.63) [lower limit 0.63]
  Part 1 - Up to 420 days post-treatment (Visit 11) | 2.27 (0.98) [lower limit 0.98] | 2.31 (1.00) [lower limit 1.00]
  Part 1 - Change from Baseline (Visit 11) | -0.47 (0.74) [lower limit 0.74] | -0.41 (0.79) [lower limit 0.79]
  Part 2 - Year 2: (FU Visit 1) | 2.5 (0.95) [lower limit 0.95] | 2.57 (0.88) [lower limit 0.88]
  Part 2 - Year 2: Change from Baseline (FU Visit 1) | -0.23 (0.87) [lower limit 0.87] | -0.17 (0.90) [lower limit 0.90]
  Part 2 - Year 3 (FU Visit 3) | 2.17 (0.98) [lower limit 0.98] | 2.25 (0.91) [lower limit 0.91]
  Part 2 - Year 3: Change from Baseline (FU Visit 3) | -0.56 (0.86) [lower limit 0.86] | -0.45 (0.87) [lower limit 0.87]
  Part 2 - Year 4 (FU Visit 5) | 2.09 (1.01) [lower limit 1.01] | 2.22 (1.00) [lower limit 1.00]
  Part 2 - Year 4: Change from Baseline (FU Visit 5) | -0.64 (0.89) [lower limit 0.89] | -0.48 (0.87) [lower limit 0.87]

12. Secondary Outcome: Part 1 - Number of Subjects With Clinical Signs/ Symptoms of Chagas Disease at Visit 1
Description: The evaluation was based on clinical examinations.
Time Frame: At Visit 1 (before treatment started)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants | 2 | 0

13. Secondary Outcome: Part 1 - Number of Subjects With Clinical Signs/ Symptoms of Chagas Disease at Visit 3
Description: The evaluation was based on clinical examinations.
Time Frame: Up to 7 days (Visit 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Anemia | 1 | 0
  Chagas disease | 2 | 0
  Hepatomegaly | 1 | 0
  Known ECG abnormality | 4 | 0

14. Secondary Outcome: Part 1 - Number of Subjects With Clinical Signs/ Symptoms of Chagas Disease at Visit 6
Description: The evaluation was based on clinical examinations.
Time Frame: Up to 30 days (Visit 6)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 215 | 110
Participants
  Known ECG abnormality | 1 | 0
  Romana sign | 0 | 1

15. Secondary Outcome: Part 1 - Number of Subjects With Clinical Signs/ Symptoms of Chagas Disease at Visit 8
Description: The evaluation was based on clinical examinations.
Time Frame: Up to 60 days (Visit 8; end of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 217 | 109
Participants
  Anemia | 1 | 0
  Chagas disease | 1 | 0
  Known ECG abnormality | 1 | 0
  Lymphadenopathy | 1 | 0

16. Secondary Outcome: Part 1 - Number of Subjects With Clinical Signs/ Symptoms of Chagas Disease at Visit 9
Description: The evaluation was based on clinical examinations.
Time Frame: Up to 90 days (Visit 9 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 213 | 107
Participants | 1 | 0

17. Secondary Outcome: Part 1 - Number of Subjects With Clinical Signs/ Symptoms of Chagas Disease at Visit 10
Description: The evaluation was based on clinical examinations.
Time Frame: Up to 240 days (Visit 10 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 212 | 109
Participants | 1 | 0

18. Secondary Outcome: Part 1 - Number of Subjects With Clinical Signs/ Symptoms of Chagas Disease at Visit 11
Description: The evaluation was based on clinical examinations.
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 210 | 108
Participants | 3 | 3

19. Secondary Outcome: Part 1 - Number of Subjects With Positive Results in Concentration Test for T. Cruzi (for Subjects <8 Months of Age)
Time Frame: Up to 90 days (Visit 9 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 12 | 7
Participants
  Visit 1|Positive | 12 | 7
  Visit 3|Positive | 1 | 1
  Visit 6|Positive | 0 | 0
  Visit 8|Positive | 0 | 0
  Visit 9|Positive | 1 | 0
  Visit 1|Negative | 0 | 0
  Visit 3|Negative | 11 | 5
  Visit 6|Negative | 12 | 7
  Visit 8|Negative | 12 | 7
  Visit 9|Negative | 11 | 7
  Visit 1|Missing | 0 | 0
  Visit 3|Missing | 0 | 1
  Visit 6|Missing | 0 | 0
  Visit 8|Missing | 0 | 0
  Visit 9|Missing | 0 | 0

20. Secondary Outcome: Part 1 - Number of Subjects With a Positive Serological Response Using Non-conventional Enzyme-linked Immunosorbent Assay-F29 (ELISAF29) Test
Description: The non-conventional ELISA-F29 test is considered an early marker of treatment efficacy in chronic Chagas disease.
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Reactive | 96 | 54
  Non-reactive | 114 | 54
  Missing | 9 | 3

21. Secondary Outcome: Part 1 - Number of Subjects With Positive Quantitative Polymerase Chain Reaction (qPCR) Results
Description: The qPCR is molecular technique, considered a tool to diagnose acute and congenital Chagas disease, as well as a marker to measure treatment failure when demonstrating positive (detectable) results
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Visit 1 - Non-detectable | 99 | 53
  Visit 1 - Detectable | 117 | 57
  Visit 1 - Non-evaluable | 1 | 1
  Visit 1 - Missing | 2 | 0
  Visit 3 - Non-detectable | 171 | 86
  Visit 3 - Detectable | 46 | 21
  Visit 3 - Non-evaluable | 0 | 1
  Visit 3 - Missing | 2 | 3
  Visit 6 - Non-detectable | 207 | 105
  Visit 6 - Detectable | 4 | 3
  Visit 6 - Non-evaluable | 3 | 2
  Visit 6 - Missing | 5 | 1
  Visit 8 - Non-detectable | 210 | 105
  Visit 8 - Detectable | 3 | 1
  Visit 8 - Non-evaluable | 2 | 2
  Visit 8 - Missing | 4 | 3
  Visit 10 - Non-detectable | 206 | 105
  Visit 10 - Detectable | 3 | 2
  Visit 10 - Non-evaluable | 2 | 2
  Visit 10 - Missing | 8 | 2
  Visit 11 - Non-detectable | 205 | 102
  Visit 11 - Detectable | 3 | 5
  Visit 11 - Non-evaluable | 1 | 1
  Visit 11 - Missing | 10 | 3

22. Secondary Outcome: Part 1 - Number of Subjects With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: TEAEs comprised events which first occurred or worsened at or after first application of study drug during the course of the study up to and including 7 days after last application of study drug
Time Frame: up to 7 days after last application of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Any treatment-emergent adverse event (TEAE) | 147 | 66
  Any Serious TEAE | 6 | 3

23. Secondary Outcome: Part 2 - Number of Subjects With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: TEAEs comprised events which first occurred or worsened at study start up to end of study in part 2.
  In Part 2, only AEs considered at least possibly related to nifurtimox (administered in part 1) and those caused by protocol-related procedures were reported.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 197 | 98
Participants
  Any AE | 0 | 0
  Any study drug-related AE | 0 | 0
  Any AE related to protocol | 0 | 0
  Any SAE | 0 | 0
  Any study drug-related SAE | 0 | 0
  Any SAE related to protocol | 0 | 0
  AE with outcome death | 0 | 0

24. Secondary Outcome: Part 1 - Number of Subjects With Treatment-emergent High Blood Chemistry Abnormalities by Treatment
Description: The Number Analyzed represents the number of subjects at baseline with a normal or lower than normal laboratory assessment who also had at least one valid laboratory value after start of treatment.
  The number of subjects represents subjects with at least one high laboratory assessment after start of treatment who had a normal or lower than normal laboratory assessment at baseline.
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Creatinine (mg/dL) | 3 | 2
  Albumin (g/dL) | 49 | 21
  Alkaline Phosphatase (U/L) | 11 | 3
  Alanine Aminotransferase (U/L) | 19 | 7
  Aspartate Aminotransferase (U/L) | 27 | 7
  Bilirubin (mg/dL) | 19 | 9
  Direct Bilirubin (mg/dL) | 21 | 9
  Blood Urea Nitrogen (mg/dL) | 11 | 3
  Urate (mg/dL) | 7 | 1
  Glucose (mg/dL) | 15 | 13
  Protein (g/dL) | 42 | 14

25. Secondary Outcome: Part 1 - Number of Subjects With Treatment-emergent Low Blood Chemistry Abnormalities by Treatment
Description: The number analyzed represents the number of subjects at baseline with a normal or higher than normal laboratory assessment who also had at least one valid laboratory value after start of treatment.
  The number of subjects represents subjects with at least one low laboratory assessment after start of treatment who had a normal or higher than normal laboratory assessment at baseline.
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Creatinine (mg/dL) | 22 | 10
  Albumin (g/dL) | 14 | 4
  Alkaline Phosphatase (U/L) | 4 | 4
  Alanine Aminotransferase (U/L) | 6 | 3
  Aspartate Aminotransferase (U/L) | 1 | 5
  Bilirubin (mg/dL) | 7 | 3
  Direct Bilirubin (mg/dL) | 0 | 0
  Blood Urea Nitrogen (mg/dL) | 31 | 15
  Urate (mg/dL) | 32 | 18
  Glucose (mg/dL) | 29 | 18
  Protein (g/dL) | 17 | 15

26. Secondary Outcome: Part 1 - Number of Subjects With Treatment-emergent High Hematology Abnormalities by Treatment
Description: The number analyzed represents the number of subjects at baseline with a normal or lower than normal laboratory assessment who also had at least one valid laboratory value after start of treatment. Subjects with missing or high abnormal values at baseline are not included in the number analyzed.
  The number of subjects represents subjects with at least one high laboratory assessment after start of treatment who had a normal or lower than normal laboratory assessment at baseline.
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Hematocrit (% | 19 | 8
  Hemoglobin (g/dL) | 15 | 3
  Erythrocytes (T/L) in Blood | 21 | 9
  Ery. Mean Corpuscular Volume (fL) in Blood | 20 | 7
  Ery. Mean Corpuscular Hemoglobin (pg) in Blood | 14 | 5
  Ery. Mean Corpuscular HGB Conc. (g/dL) in Blood | 23 | 6
  Leukocytes (GIGA/L) in Blood | 41 | 16
  Neutrophils/Leukocytes (%) | 38 | 12
  Neutrophils (GIGA/L) | 36 | 8
  Lymphocytes/Leukocytes (%) | 35 | 17
  Lymphocytes (GIGA/L) | 21 | 7
  Monocytes/Leukocytes (%) | 33 | 17
  Monocytes (GIGA/L) | 17 | 15
  Eosinophils/Leukocytes (%) | 58 | 26
  Eosinophils (GIGA/L) | 53 | 22
  Basophils/Leukocytes (%) | 20 | 7
  Basophils (GIGA/L) | 10 | 2
  Platelets (GIGA/L) in Blood | 27 | 13

27. Secondary Outcome: Part 1 - Number of Subjects With Treatment-emergent Low Hematology Abnormalities by Treatment
Description: The number analyzed represents the number of subjects at baseline with a normal or lower than normal laboratory assessment who also had at least one valid laboratory value after start of treatment. Subjects with missing or low abnormal values at baseline are not included in the number analyzed.
  The number of subjects represents subjects with at least one low laboratory assessment after start of treatment who had a normal or higher than normal laboratory assessment at baseline.
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Hematocrit (% | 30 | 17
  Hemoglobin (g/dL) | 23 | 17
  Erythrocytes (T/L) in Blood | 15 | 9
  Ery. Mean Corpuscular Volume (fL) in Blood | 16 | 6
  Ery. Mean Corpuscular Hemoglobin (pg) in Blood | 19 | 10
  Ery. Mean Corpuscular HGB Conc. (g/dL) in Blood | 29 | 21
  Leukocytes (GIGA/L) in Blood | 39 | 18
  Neutrophils/Leukocytes (%) | 53 | 27
  Neutrophils (GIGA/L) | 46 | 25
  Lymphocytes/Leukocytes (%) | 40 | 9
  Lymphocytes (GIGA/L) | 5 | 0
  Monocytes/Leukocytes (%) | 54 | 28
  Monocytes (GIGA/L) | 33 | 22
  Eosinophils/Leukocytes (%) | 13 | 5
  Eosinophils (GIGA/L) | 14 | 5
  Basophils/Leukocytes (%) | 1 | 2
  Basophils (GIGA/L) | 1 | 2
  Platelets (GIGA/L) in Blood | 6 | 3

28. Secondary Outcome: Part 1 - Number of Subjects With Treatment-emergent High Coagulation Abnormalities by Treatment
Description: as for outcome 24
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Prothrombin Time (sec) in Plasma | 38 | 23
  Activated Partial Thromboplastin | 9 | 10
  Time in Plasma Prothrombin Intl. Normalized Ratio | 21 | 13

29. Secondary Outcome: Part 1 - Number of Subjects With Treatment-emergent Low Coagulation Abnormalities by Treatment
Description: as for outcome 25
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants
  Prothrombin Time (sec) in Plasma | 10 | 5
  Activated Partial Thromboplastin | 15 | 2
  Time in Plasma Prothrombin Intl. Normalized Ratio | 14 | 5

30. Secondary Outcome: Part 1 - Number of Subjects With Abnormal Urinalysis Findings Considered as Clinically Significant or Reported as Adverse Events (AEs)
Description: Urinalysis was performed and the following parameters evaluated: bilirubin, blood (red blood cells, white blood cells), chorionic gonadotropin β, glucose, ketones, leukocytes, nitrite, pH, protein, specific gravity, and urobilinogen.
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants | 0 | 0

31. Secondary Outcome: Part 1 - Number of Subjects With Abnormal ECG Findings Considered as Clinically Significant by Investigators
Description: Clinical significance of abnormal ECG was based on the judgement of the investigator
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
Participants | 0 | 0

32. Secondary Outcome: Part 1 - Mean Changes in Vital Signs (Systolic Blood Pressure) Between the Treatment Groups From Baseline
Description: Systolic Blood Pressure
Time Frame: Baseline and up to 420 days (Visit 11 post-treatment)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
mmHg
  VISIT 1 | 1.09 (7.79) [lower limit 7.79] | 0.69 (7.85) [lower limit 7.85]
  VISIT 2 | -3.75 (7.50) [lower limit 7.50] | -5.00 (7.07) [lower limit 7.07]
  VISIT 3 | 1.08 (9.98) [lower limit 9.98] | -0.50 (8.45) [lower limit 8.45]
  VISIT 6 | -0.74 (10.70) [lower limit 10.70] | -1.12 (9.89) [lower limit 9.89]
  VISIT 8 | -0.41 (11.01) [lower limit 11.01] | 0.48 (11.24) [lower limit 11.24]
  VISIT 9 | -0.13 (11.11) [lower limit 11.11] | -0.45 (10.49) [lower limit 10.49]
  VISIT 10 | -0.02 (10.46) [lower limit 10.46] | -1.48 (10.95) [lower limit 10.95]
  VISIT 11 | 1.20 (11.52) [lower limit 11.52] | 1.57 (10.70) [lower limit 10.70]

33. Secondary Outcome: Part 1 - Mean Changes in Vital Signs (Diastolic Blood Pressure) Between the Treatment Groups From Baseline
Description: Diastolic Blood Pressure
Time Frame: Baseline and up to 420 days (Visit 11 post-treatment)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
mmHg
  VISIT 1 | 1.00 (7.72) [lower limit 7.72] | 0.90 (7.90) [lower limit 7.90]
  VISIT 2 | -1.25 (2.50) [lower limit 2.50] | -1.00 (2.00) [lower limit 2.00]
  VISIT 3 | 0.76 (8.36) [lower limit 8.36] | 0.26 (8.05) [lower limit 8.05]
  VISIT 6 | 0.26 (10.87) [lower limit 10.87] | -0.14 (10.21) [lower limit 10.21]
  VISIT 8 | 0.08 (9.91) [lower limit 9.91] | 0.93 (10.17) [lower limit 10.17]
  VISIT 9 | -0.68 (8.81) [lower limit 8.81] | -0.21 (10.03) [lower limit 10.03]
  VISIT 10 | 0.99 (9.90) [lower limit 9.90] | 0.85 (9.53) [lower limit 9.53]
  VISIT 11 | 2.30 (11.06) [lower limit 11.06] | 3.25 (10.95) [lower limit 10.95]

34. Secondary Outcome: Part 1 - Mean Changes in Vital Signs (Respiratory Rate) Between the Treatment Groups From Baseline
Description: Respiratory Rate
Time Frame: Baseline and up to 420 days (Visit 11 post-treatment)
Measure: Mean (Standard Deviation); unit: BREATHS/MIN
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
BREATHS/MIN
  VISIT 1 | 0.12 (4.10) [lower limit 4.10] | 0.47 (2.91) [lower limit 2.91]
  VISIT 2 | -1.50 (3.42) [lower limit 3.42] | -1.00 (1.15) [lower limit 1.15]
  VISIT 3 | -0.05 (3.15) [lower limit 3.15] | -0.14 (3.91) [lower limit 3.91]
  VISIT 6 | -0.57 (4.16) [lower limit 4.16] | -0.06 (3.87) [lower limit 3.87]
  VISIT 8 | -0.77 (4.04) [lower limit 4.04] | 0.04 (4.58) [lower limit 4.58]
  VISIT 9 | -1.01 (4.06) [lower limit 4.06] | -0.50 (3.76) [lower limit 3.76]
  VISIT 10 | -1.36 (4.50) [lower limit 4.50] | -0.24 (3.60) [lower limit 3.60]
  VISIT 11 | -1.93 (5.10) [lower limit 5.10] | -0.74 (4.61) [lower limit 4.61]

35. Secondary Outcome: Part 1 - Mean Changes in Vital Signs (Heart Rate) Between the Treatment Groups From Baseline
Description: Heart Rate
Time Frame: Baseline and up to 420 days (Visit 11 post-treatment)
Measure: Mean (Standard Deviation); unit: BEATS/MIN
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
BEATS/MIN
  VISIT 1 | -1.08 (10.19) [lower limit 10.19] | 0.26 (11.37) [lower limit 11.37]
  VISIT 2 | -6.75 (2.22) [lower limit 2.22] | -0.75 (2.99) [lower limit 2.99]
  VISIT 3 | 0.04 (10.11) [lower limit 10.11] | -0.51 (11.46) [lower limit 11.46]
  VISIT 6 | -0.78 (11.49) [lower limit 11.49] | -0.75 (11.92) [lower limit 11.92]
  VISIT 8 | -1.27 (11.65) [lower limit 11.65] | -1.34 (11.03) [lower limit 11.03]
  VISIT 9 | -1.26 (11.97) [lower limit 11.97] | -1.63 (10.56) [lower limit 10.56]
  VISIT 10 | -3.28 (11.87) [lower limit 11.87] | -3.28 (11.61) [lower limit 11.61]
  VISIT 11 | -3.57 (12.57) [lower limit 12.57] | -4.66 (14.73) [lower limit 14.73]

36. Secondary Outcome: Part 1 - Mean Changes in Vital Signs (Body Temperature) Between the Treatment Groups From Baseline
Description: Temperature
Time Frame: Baseline and up to 420 days (Visit 11 post-treatment)
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Nifurtimox 60 Days / Arm 1 | Nifurtimox 30 Days, Then Placebo 30 Days / Arm 2
Number analyzed (Participants) | 219 | 111
°C
  VISIT 1 | 0.01 (0.39) [lower limit 0.39] | 0.04 (0.36) [lower limit 0.36]
  VISIT 2 | -0.35 (0.45) [lower limit 0.45] | -0.03 (0.39) [lower limit 0.39]
  VISIT 3 | -0.10 (0.36) [lower limit 0.36] | 0.04 (0.43) [lower limit 0.43]
  VISIT 6 | -0.06 (0.44) [lower limit 0.44] | 0 (0.44) [lower limit 0.44]
  VISIT 8 | -0.06 (0.45) [lower limit 0.45] | 0.05 (0.42) [lower limit 0.42]
  VISIT 9 | -0.03 (0.44) [lower limit 0.44] | 0.02 (0.47) [lower limit 0.47]
  VISIT 10 | -0.07 (0.49) [lower limit 0.49] | -0.01 (0.52) [lower limit 0.52]
  VISIT 11 | -0.14 (0.51) [lower limit 0.51] | -0.10 (0.50) [lower limit 0.50]

37. Other Pre Specified Outcome: Part 1: Number of Participants Cured With 60-day Regimen Compared With Historical Active Control (Benznidazole)
Description: This exploratory efficacy analysis evaluated the cure rate assessed as seroconversion of nifurtimox after 1-year post-treatment follow-up with that of published data for benznidazole (Sosa Estani et al. 1998 and de Andrade et al. 1996) at 4- and 3-year post-treatment follow-up, respectively, used as historical control.
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox 60 Days / Arm 1
Number analyzed (Participants) | 219
Participants | 10

38. Other Pre Specified Outcome: Part 1 - Relationship of Conventional Serology (Total Purified Antigen ELISA) and qPCR Testing by Visit
Description: Using frequencies of matches and mismatches to assess agreement
  Reactive = Reac ELISA Detectable = Detec qPCR Non-reactive = Nonreac ELISA Non-detectable = Nondetec qPCR Non evaluable = Noneval qPCR qPCR Missing = Miss qPCR Missing conventional testing = Miss ELISA
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Nifurtimox 60 Days Reactive Detectable: Nifurtimox 60 days with Reac ELISA and Detec qPCR
- Nifurtimox 60 Days Reactive Non-detectable: Nifurtimox 60 days with Reac ELISA and Nondetec qPCR
- Nifurtimox 60 Days Non-reactive Detectable: Nifurtimox 60 days with Nonreac ELISA and Detec qPCR
- Nifurtimox 60 Days Non-reactive Non-detectable: Nifurtimox 60 days with Nonreac ELISA and Nondetec qPCR
- Nifurtimox 60 Days Reactive Non Evaluable: Nifurtimox 60 days with Reac ELISA and Non evaluable qPCR
- Nifurtimox 60 Days Reactive qPCR Missing: Nifurtimox 60 days with Reac ELISA and missing qPCR
- Nifurtimox 30 Days Reactive Detectable: Nifurtimox 30 days with Reac ELISA and Detec qPCR
- Nifurtimox 30 Days Reactive Non-detectable: Nifurtimox 30 days with Reac ELISA and Nondetec qPCR
- Nifurtimox 30 Days Non-reactive Detectable: Nifurtimox 30 days with Nonreac ELISA and Detec qPCR
- Nifurtimox 30 Days Non-reactive Non-detectable: Nifurtimox 30 days with Nonreac ELISA and Nondetec qPCR
- Nifurtimox 30 Days Reactive Non Evaluable: Nifurtimox 30 days with Reac ELISA and Non evaluable qPCR
- Nifurtimox 30 Days Missing Conventional Testing Non-detectable: Nifurtimox 30 days with Miss ELISA and Nondetec qPCR
Arm/Group | Nifurtimox 60 Days Reactive Detectable | Nifurtimox 60 Days Reactive Non-detectable | Nifurtimox 60 Days Non-reactive Detectable | Nifurtimox 60 Days Non-reactive Non-detectable | Nifurtimox 60 Days Reactive Non Evaluable | Nifurtimox 60 Days Reactive qPCR Missing | Nifurtimox 30 Days Reactive Detectable | Nifurtimox 30 Days Reactive Non-detectable | Nifurtimox 30 Days Non-reactive Detectable | Nifurtimox 30 Days Non-reactive Non-detectable | Nifurtimox 30 Days Reactive Non Evaluable | Nifurtimox 30 Days Missing Conventional Testing Non-detectable
Number analyzed (Participants) | 219 | 219 | 219 | 219 | 219 | 219 | 111 | 111 | 111 | 111 | 111 | 111
Participants
  Visit 1 | 117 | 99 | 0 | 0 | 1 | 2 | 57 | 52 | 0 | 1 | 1 | 0
  Visit 8 | 3 | 210 | 0 | 0 | 2 | 0 | 1 | 103 | 0 | 1 | 2 | 1
  Visit 10 | 3 | 195 | 0 | 11 | 2 | 0 | 2 | 99 | 0 | 6 | 2 | 0
  Visit 11 | 3 | 194 | 0 | 11 | 1 | 1 | 5 | 96 | 0 | 6 | 1 | 0

39. Other Pre Specified Outcome: Part 1 - Relationship of Conventional Serology (Total Purified Antigen ELISA) and Non-conventional (ELISA-F29) Serologic Testing by Visit
Description: Using frequencies of matches and mismatches to assess agreement
  Reactive = Reac ELISA Reactive = Reac F29 Non-reactive = Nonreac ELISA Non-reactive = Nonreac F29
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Nifurtimox 60 Days Reactive and Reactive: Nifurtimox 60 days with Reac ELISA and Reac F29
- Nifurtimox 60 Days Reactive and Non-reactive: Nifurtimox 60 days with Reac ELISA and Nonreac F29
- Nifurtimox 60 Days Non-reactive and Reactive: Nifurtimox 60 days with Nonreac ELISA and Reac F29
- Nifurtimox 60 Days Non-reactive and Non-reactive: Nifurtimox 60 days with Nonreac ELISA and Nonreac F29
- Nifurtimox 30 Days Reactive and Reactive: Nifurtimox 30 days with Reac ELISA and Reac F29
- Nifurtimox 30 Days Reactive and Non-reactive: Nifurtimox 30 days with Reac ELISA and Nonreac F29
- Nifurtimox 30 Days Non-reactive and Reactive: Nifurtimox 30 days with Nonreac ELISA and Reac F29g
- Nifurtimox 30 Days Non-reactive and Non-reactive: Nifurtimox 30 days Nonreac ELISA and Nonreac F29
Arm/Group | Nifurtimox 60 Days Reactive and Reactive | Nifurtimox 60 Days Reactive and Non-reactive | Nifurtimox 60 Days Non-reactive and Reactive | Nifurtimox 60 Days Non-reactive and Non-reactive | Nifurtimox 30 Days Reactive and Reactive | Nifurtimox 30 Days Reactive and Non-reactive | Nifurtimox 30 Days Non-reactive and Reactive | Nifurtimox 30 Days Non-reactive and Non-reactive
Number analyzed (Participants) | 219 | 219 | 219 | 219 | 111 | 111 | 111 | 111
Participants
  Visit 1 | 142 | 77 | 0 | 0 | 72 | 38 | 0 | 1
  Visit 3 | 133 | 85 | 0 | 0 | 64 | 43 | 0 | 1
  Visit 6 | 131 | 83 | 0 | 0 | 67 | 42 | 0 | 1
  Visit 8 | 124 | 91 | 0 | 63 | 63 | 43 | 0 | 1
  Visit 10 | 108 | 92 | 2 | 9 | 61 | 42 | 0 | 6
  Visit 11 | 93 | 106 | 3 | 8 | 54 | 48 | 0 | 6

40. Other Pre Specified Outcome: Part 1 - Relationship of Conventional Serology (Recombinant ELISA) and Non-conventional (ELISA-F29) Serologic Testing by Visit
Description: Using frequencies of matches and mismatches to assess agreement
  Reactive = Reac ELISA Reactive = Reac F29 Non-reactive = Nonreac ELISA Non-reactive= Nonreac F29
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Nifurtimox 60 Days Reactive and Reactive: Nifurtimox 60 days Reac ELISA and Reac F29
- Nifurtimox 60 Days Non-reactive and Non-reactive: Nifurtimox 60 days Nonreac ELISA and Nonreac F29
- Nifurtimox 30 Days Reactive and Reactive: Nifurtimox 30 days with Reactive ConvReac ELISA and Reac F29
- Nifurtimox 30 Days Non-reactive and Reactive: Nifurtimox 30 days with Nonreac ELISA and Reac F29
- Nifurtimox 30 Days Non-reactive and Non-reactive: Nifurtimox 30 days with Nonreac ELISA and Nonreac F29
Arm/Group | Nifurtimox 60 Days Reactive and Reactive | Nifurtimox 60 Days Reactive and Non-reactive | Nifurtimox 60 Days Non-reactive and Reactive | Nifurtimox 60 Days Non-reactive and Non-reactive | Nifurtimox 30 Days Reactive and Reactive | Nifurtimox 30 Days Non-reactive and Reactive | Nifurtimox 30 Days Non-reactive and Non-reactive
Number analyzed (Participants) | 219 | 219 | 219 | 219 | 111 | 111 | 111
Participants
  Visit 1 | 142 | 77 | 0 | 0 | 72 | 0 | 1
  Visit 3 | 133 | 85 | 0 | 0 | 64 | 0 | 1
  Visit 6 | 131 | 81 | 0 | 2 | 67 | 0 | 1
  Visit 8 | 124 | 90 | 0 | 1 | 63 | 0 | 1
  Visit 10 | 108 | 91 | 2 | 10 | 59 | 2 | 5
  Visit 11 | 93 | 106 | 3 | 0 | 53 | 1 | 6

41. Other Pre Specified Outcome: Part 1 - Relationship of Conventional Serology (ELISA) to Indirect Hemagglutination Assay (IHA) Results
Description: Sero-reduction is defined as a => 20% reduction in optical density [OD]) using two conventional ELISA serology tests in subjects => 8 months to < 18 years of age at randomization; Others: reactive results that are not sero-reduction in subjects => 8 months to < 18 years of age at randomization; or reactive results in subjects < 8 months of age at randomization.
  Non-reactive ELISA = Nonreac ELISA Non-reactive IHA = Nonreac IHA Reactive IHA decrease = Reac IHA dec React IHA nochange = Reac IHA nochange Reactive ELISA: seroreduction = Reac ELISA reduc Reactive ELISA: others = Reac ELISA other
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Non-reactive ELISA and Non-reactive IHA: Nonreac ELISA and Nonreac IHA
- Non-reactive ELISA and Reactive IHA Decrease: Nonreac ELISA and Reac IHA dec
- Non-react ELISA and React IHA Nochange: Nonreac ELISA and Reac IHA nochange
- Reactive ELISA: Sero-reduction and Non-react IHA: Reac ELISA and Nonreac IHA
- Reactive ELISA: Sero Reduction and Reactive IHA Decrease: Reac ELISA reduc and Reac IHA dec
- Reactive ELISA: Sero-reduction and Reactive IHA Nochange: Reac ELISA reduc and Reac IHA nochange
- Reactive ELISA: Others and Non-reactive IHA: Reac ELISA other and Nonreac IHA
- Reactive ELISA: Others and React IHA Decrease: Reac ELISA other and Reac IHA dec
- Reactive ELISA: Others and React IHA Nochange: Reac ELISA other and Reac IHA nochange
- Reactive ELISA: Others and Missing IHA: Reac ELISA other and IHA missing
Arm/Group | Non-reactive ELISA and Non-reactive IHA | Non-reactive ELISA and Reactive IHA Decrease | Non-react ELISA and React IHA Nochange | Reactive ELISA: Sero-reduction and Non-react IHA | Reactive ELISA: Sero Reduction and Reactive IHA Decrease | Reactive ELISA: Sero-reduction and Reactive IHA Nochange | Reactive ELISA: Others and Non-reactive IHA | Reactive ELISA: Others and React IHA Decrease | Reactive ELISA: Others and React IHA Nochange | Reactive ELISA: Others and Missing IHA
Number analyzed (Participants) | 318 | 318 | 318 | 318 | 318 | 330 | 318 | 318 | 318 | 318
Participants
  Nifurtimox 60 days | 8 | 2 | 0 | 2 | 40 | 20 | 1 | 47 | 89 | 1
  Nifurtimox 30 days | 4 | 1 | 0 | 0 | 12 | 4 | 1 | 30 | 58 | 0

42. Other Pre Specified Outcome: Part 1 - Relationship Between Conventional ELISA Results in Terms of Cure or No Cure and IHA Results in All Patients
Description: Cure is defined as sero-reduction (in subjects => 8 months to < 18 years of age at randomization) or sero-conversion (in all subjects). Sero-reduction is defined as a => 20% reduction in optical density [OD]) measured by two conventional ELISA serology tests and sero-conversion is defined as negative Immunoglobulin G [IgG] concentration measured by two conventional ELISA serology tests.
  Cure = Cure Non reactive/reactive decreasing = Nonreac/reac dec Reactive non-decreasing = Reac nondec No cure = No Cure Missing IHA testing = IHA missing
Time Frame: Up to 420 days (Visit 11 post-treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Cure and Non Reactive/Reactive Decreasing: ELISA Cure and IHA Nonreac/reac dec
- Cure and Reactive Non-decreasing: ELISA Cure and IHA Reac nondec
- No Cure and Non Reactive/Reactive Decreasing: ELISA No Cure and IHA results: Nonreac/reac dec
- No Cure and Reactive Non-decreasing: ELISA No Cure and IHA Reac nondec
- No Cure and Missing IHA Testing: ELISA No Cure and IHA missing
Arm/Group | Cure and Non Reactive/Reactive Decreasing | Cure and Reactive Non-decreasing | No Cure and Non Reactive/Reactive Decreasing | No Cure and Reactive Non-decreasing | No Cure and Missing IHA Testing
Number analyzed (Participants) | 318 | 318 | 318 | 318 | 318
Participants
  Nifurtimox 60 days | 52 | 20 | 48 | 89 | 1
  Nifurtimox 30 days | 17 | 4 | 29 | 58 | 0

ADVERSE EVENTS:
Time Frame: Part 1: From first application of study drug up to and including 7 days after last application of study drug Part 2: first occurred or worsened at start of study part 2 up to 3 years.
Groups:
- Nifurtimox 60-day Regimen: Nifurtimox daily dose 8-10 mg/kg (adolescents, 40-60 kg) or 10-20 mg/kg (infants/children, below 40 kg) for 60 days
- Nifurtimox 30-day Regimen: Nifurtimox daily dose 8-10 mg/kg (adolescents, 40-60 kg) or 10-20 mg/kg (infants/children, below 40 kg) for 30 days followed by placebo
Arm/Group | Nifurtimox 60-day Regimen | Nifurtimox 30-day Regimen
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/111
Serious Adverse Events (participants affected / at risk) | 6/219 | 3/111
Other Adverse Events (participants affected / at risk) | 128/219 | 51/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nifurtimox 60-day Regimen (N=219) | Nifurtimox 30-day Regimen (N=111)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nifurtimox 60-day Regimen (N=219) | Nifurtimox 30-day Regimen (N=111)
Abdominal pain (Gastrointestinal disorders) | 19 (27) | 9 (11)
Abdominal pain upper (Gastrointestinal disorders) | 15 (20) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 16 (17) | 6 (7)
Nausea (Gastrointestinal disorders) | 19 (24) | 14 (15)
Vomiting (Gastrointestinal disorders) | 33 (57) | 10 (11)
Pyrexia (General disorders) | 20 (25) | 4 (5)
Bronchitis (Infections and infestations) | 12 (14) | 6 (7)
Nasopharyngitis (Infections and infestations) | 22 (28) | 11 (13)
Pharyngitis (Infections and infestations) | 13 (13) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 13 (17) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 25 (27) | 8 (8)
Headache (Nervous system disorders) | 30 (44) | 16 (23)

LIMITATIONS AND CAVEATS:
Abnormal findings on neurological examination by physical examination after Screening will be documented as AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT02625974/Prot_002.pdf
  • Statistical Analysis Plan (2020-01-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT02625974/SAP_003.pdf